CLINICAL TRIAL: NCT07070544
Title: Head of Department of Physical Therapy for Cardiovascular/Respiratory Disorders and Geriatrics
Brief Title: Effect of Electromagnetic Field Therapy and Customized Foot Insole on Peripheral Circulation and Ankle-Brachial Pressure Index in Patients With Diabetic Foot Ulcer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Ibrahim ismail Abuzaid, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: South Valley University PTh
Record Dates: First submitted 2025-06-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Diabetic Foot Ulcer
Keywords: Effect of Electromagnetic Field Therapy; Customized Foot Insole; Peripheral Circulation; Ankle-Brachial Pressure Index
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study Group (Active Comparator): Electromagnetic Field Therapy:
  * Frequency: 50 Hz
  * Intensity: 5-30 mT
  * Duration: 30 minutes/session
  * Frequency: 3 sessions/week for 8 weeks
  Customized Foot Insoles:
  * Individually tailored based on foot pressure mapping and deformity.
  * Designed to offload pressure points and support foot arches.
  Standard Care:
  • Wound care, glycemic control, and patient education as per institutional protocol.
  Interventions: Device: Electromagnetic Field Therapy: • Frequency: 50 Hz • Intensity: 5-30 mT • Duration: 30 minutes/session • Frequency: 3 sessions/week for 8 weeks Customized Foot Insoles: • Individually tailored based on
- The control group (Placebo Comparator): Standard Care:
  • Wound care, glycemic control, and patient education as per institutional protocol.
  Interventions: Device: Electromagnetic Field Therapy: • Frequency: 50 Hz • Intensity: 5-30 mT • Duration: 30 minutes/session • Frequency: 3 sessions/week for 8 weeks Customized Foot Insoles: • Individually tailored based on

INTERVENTIONS:
Device: Electromagnetic Field Therapy: • Frequency: 50 Hz • Intensity: 5-30 mT • Duration: 30 minutes/session • Frequency: 3 sessions/week for 8 weeks Customized Foot Insoles: • Individually tailored based on — Electromagnetic Field Therapy:
  * Frequency: 50 Hz
  * Intensity: 5-30 mT
  * Duration: 30 minutes/session
  * Frequency: 3 sessions/week for 8 weeks
  Customized Foot Insoles:
  * Individually tailored based on foot pressure mapping and deformity.
  * Designed to offload pressure points and support foot arches.
  Standard Care:
  • Wound care, glycemic control, and patient education as per institutional protocol.

SUMMARY:
Diabetic foot ulcers (DFUs) are a significant complication of diabetes mellitus, associated with poor peripheral circulation, neuropathy, and increased risk of lower-limb amputation. Optimizing peripheral blood flow is critical in the prevention and management of DFUs. Traditional offloading strategies, such as customized foot insoles, have demonstrated efficacy in reducing plantar pressure and promoting ulcer healing.

Electromagnetic field (EMF) therapy is a non-invasive modality that has shown potential in enhancing microcirculation, promoting angiogenesis, and modulating inflammatory processes. Preliminary studies have suggested that EMF may improve peripheral circulation and tissue oxygenation in diabetic patients.

This study aims to investigate the combined effect of EMF therapy and customized foot insoles on peripheral circulation and Ankle-Brachial Pressure Index (ABPI) in patients with diabetic foot ulcers, hypothesizing that this integrated approach may yield superior outcomes compared to standard care.

DETAILED DESCRIPTION:
2. Objectives

Primary Objective:

• To evaluate the effect of EMF therapy combined with customized foot insoles on peripheral circulation in patients with diabetic foot ulcers.

Secondary Objective:

* To assess changes in Ankle-Brachial Pressure Index (ABPI) following intervention.
* To compare the ulcer healing rates and pain levels between intervention and control groups.

  3. Research Questions
  1. Does the combination of EMF therapy and customized foot insoles improve peripheral circulation in patients with diabetic foot ulcers?
  2. Is there a significant improvement in ABPI in the intervention group compared to control?
  3. What is the effect of the intervention on ulcer healing rates and pain reduction?

     ________________________________________
  4. Hypotheses
* H1: EMF therapy combined with customized foot insoles significantly improves peripheral circulation compared to standard care.
* H2: EMF therapy combined with customized foot insoles significantly improves ABPI in patients with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with Type 2 Diabetes Mellitus.

  * Presence of unilateral or bilateral diabetic foot ulcer.
  * ABPI between 0.6 - 1.0 (mild to moderate arterial insufficiency).

Exclusion Criteria:

* • Severe peripheral arterial disease (ABPI <0.5).

  * Active infection requiring hospitalization.
  * History of amputation.
  * Cardiac pacemaker or contraindication to EMF therapy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood flow | Measurement Timeline: • Minimum value (Baseline)(Week 0) • Mid-intervention (Week 4) • Maximum value (Post-intervention) (Week 8) • Follow-up (Week 12)
  Primary Outcome:
  • Peripheral Circulation: Assessed by Laser Doppler Flowmetry and/or skin perfusion pressure (SPP).

SECONDARY OUTCOMES:
• Ankle-Brachial Pressure Index (ABPI) | Measurement Timeline: • Minimum value (Baseline) (Week 0) • Mid-intervention (Week 4) • Maximum value (Post-intervention) (Week 8) • Follow-up (Week 12)
  • Ankle-Brachial Pressure Index (ABPI): Measured using handheld Doppler.
• Ulcer Healing Rate | Measurement Timeline: • Minimum value (Baseline) (Week 0) • Mid-intervention (Week 4) • Maximum value (Post-intervention) (Week 8) • Follow-up (Week 12)
  • Ulcer Healing Rate: Monitored through ulcer size reduction (planimetric tracing and digital photography).
• Pain Level: | Measurement Timeline: • Minimum value (Baseline) (Week 0) • Mid-intervention (Week 4) • Maximum value (Post-intervention) (Week 8) • Follow-up (Week 12)
  • Pain Level: Measured using the Visual Analog Scale (VAS).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burhan A, Arofiati F, Da Silva VA, Sebayang SM. Effect of Ankle Brachial Index (ABI) and Compression Therapy on Diabetic Foot Ulcer Healing. Curr Diabetes Rev. 2024;20(1):e310323215277. doi: 10.2174/1573399819666230331083420. PMID 37005544
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37005544/